CLINICAL TRIAL: NCT05656651
Title: ACTIVE- Acute Effects of a Single Physical Exercise Intervention on Immune Cells and Inflammation in Cancer Patients and a Healthy Comparison Group
Brief Title: Acute Immunological Effects of Exercise in Cancer Patients
Acronym: ACTIVE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Miriam Götte, Principal Investigator, Universität Duisburg-Essen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ACTIVE
Record Dates: First submitted 2022-11-13; First posted 2022-12-19 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cancer patients (Experimental): Single exercise intervention following a HIIT protocol, duration ~20 mins
  Interventions: Behavioral: High intensity interval exercise training
- Healthy adults (Active Comparator): Single exercise intervention following a HIIT protocol, duration ~20 mins
  Interventions: Behavioral: High intensity interval exercise training

INTERVENTIONS:
Behavioral: High intensity interval exercise training — Endurance training adapted to age, resting heart rate
  Other Names: HIIT, Exercise

SUMMARY:
The aim of the study is to evaluate and compare immune response to a single exercise intervention in cancer patients and healthy age-maged individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents and young adults >14 years of age
* undergoing acute cancer treatment (chemotherapy)
* signed informed consent

Exclusion Criteria:

* Inability to follow and implement test instructions
* medical contraindication to HIIT on cycle ergometer
* chemotherapeutic treatment 48 h prior
* Hb <8g/dl; platelets < 20,000/ul.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12-19 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Number of Natural Killer Cells | Change from pre Intervention to immediately after intervention and 1 hour post intervention
  NK cells, subgroups and innate lymphoid cells

SECONDARY OUTCOMES:
Subjective Quality of Life | Once after intervention
  Quality of Life (EORTC QLQ-C30, questionnaire score from 0 - 100, higher score = better quality of life)
Fatigue | Once after intervention
  Fatigue (EORTC QLQ FA12 Fatigue questionnaire range 0 - 100, higher score = worse outcome)
Nutritional status | Once after intervention
  Mini Nutritional Assessment (MNA range 0 - 14 points), lower score = worse

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Götte, Dr., Principal Investigator — University Hospital, Essen
Locations (1):
- University Hospital Essen, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Deppe I, Beller R, Kiehl F, Lazzari N, Bennstein SB, Reinhardt D, Dirksen U, Gotte M. The impact of a single HIIT intervention on the mobilization of NK cells and ILCs in adolescents and young adults (AYA) undergoing cancer treatment: an interventional controlled trial. BMC Cancer. 2025 Apr 14;25(1):689. doi: 10.1186/s12885-025-14058-3. PMID 40229731